CLINICAL TRIAL: NCT06621875
Title: Effect Of The Presence Of Dynapenia On Posture, Spine Muscle Elasticity, Strength And Endurance In Young Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Aynur Ayazzade (Other)
Responsible Party: Sponsor-Investigator, Aynur Ayazzade, Graduate Student, Atılım University
Organization: Atılım University (Other)
Other Study IDs: ATU-FTR-AY-01
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Dynapenia; Muscle Weakness; Sarcopenia
Keywords: Muscle strength; Sarcopenia; Posture; Muscle elasticity; Muscle endurance; Dynapenia; Hand Grip
MeSH Terms: conditions — Muscle Weakness; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dynapenia Group: Those with no decrease in muscle mass but decreased muscle strength and/or performance will be included in the 'dynapenia group'.
- Control Group: Those with no decrease in muscle mass, muscle function and performance will be included in the 'control group'.

SUMMARY:
The aim of the present study was to determine the effect of dynapenia on posture, spinal muscle elasticity, strength and endurance in young adults.

DETAILED DESCRIPTION:
Skeletal muscle plays an important role in general health and physical development throughout the life cycle [1]. Skeletal muscle strength and performance are of critical importance in performing daily activities, maintaining mobility, and maintaining general health. Therefore, changes in general muscle strength and performance due to various reasons differentiate muscle contraction quality and neural activation, facilitating for the concept of 'dynapenia' [2,3].

Dynapenia is defined as a decrease in performance and/or strength without loss of muscle mass [4]. Although dynapenia, which facilitates for morbidity and mortality [5,7], is a well-defined condition in the elderly, there is very limited information about its prevalence and causes in young people [8]. Dynapenia, which has many negative effects on quality of life and daily functioning for the general population [9], is considered a form of accelerated muscle aging and can be defined as the "pre-sarcopenia stage" [10].

When other causes of dynapenia are examined in the literature; age and chronic diseases have been emphasized, but it has been overlooked that one of the most important modifiable factors, inadequate physical activity, can facilitate for dynapenia, especially in young people [4]. The COVID-19 pandemic that started in 2020 and the quarantine and similar measures taken subsequently have led to a decrease in physical activity levels in young people and an increase of approximately 28% in daily sitting time [11]. Low physical activity levels and the resulting decrease in muscle strength and performance can facilitate for dynapenia in young individuals [4,12].

Individuals who spend a long time in front of the computer also struggle with many health problems caused by being inactive for a long time, especially in the neck and waist [13,14]. Posture that is disrupted by the side effects of sitting for a long time can cause a decrease in muscle length and/or elasticity in certain groups of muscles [15]. Changes in the muscle also lead to a decrease in muscle strength over time [16,17], which can be an accelerating factor for dynapenia.

In the literature, many studies have addressed postural disorders, spinal muscle elasticity, muscle strength and endurance with the functional strength parameter handgrip strength [18,21], but no study has examined these parameters in young individuals with dynapenia. When deciding on the presence of dynapenia, handgrip strength is the most important parameter that provides information about general muscle strength. However, changes in the spine in individuals with dynapenia, whose handgrip strength and general muscle performance are reduced, have been ignored in the literature.

Evaluating posture, spinal muscle strength, elasticity and endurance in individuals with dynapenia can be a fundamental step in preparing preventive and therapeutic algorithms against dynapenia. The strength and endurance of spinal muscles can play a critical role in providing postural control, preserving movement functions and reducing the risk of injury, especially in individuals with dynapenia. Therefore, examining factors related to the spine in the presence of dynapenia in young individuals can make significant contributions to developing preventive health strategies, increasing functional capacities and improving quality of life.

According to above information; The aim of the present study was to determine the effect of dynapenia on posture, spinal muscle elasticity, strength and endurance in young adults.

Data collection will be carried out as follows: Participants' height, weight, body mass index and smoking, average time spent in front of the screen during the day (hours of daily use x years of use), presence of Covid-19, number of cases and when it occurred will be recorded verbally. Physical activity level will be assessed with the International Physical Activity Questionnaire - Short Form (IPAQ-SF) [22,23]; average smartphone usage time with the Smartphone Addiction Scale Short Form [24], and sleep quality (Pittsburgh Sleep Quality Index) [25]. Those with no decrease in muscle mass but a decrease in muscle strength and/or performance will be included in the 'dypenia group', and those with no decrease in muscle mass, muscle function and performance will be included in the 'control group'.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Filling out all the survey questions

Exclusion Criteria:

* Presence of chronic diseases that may affect the musculoskeletal system (diabetes, heart disease, neurological disorders)
* Use of medications that may affect muscle functions (corticosteroids, muscle relaxants)
* Presence of serious musculoskeletal injury within the last six months
* Presence of surgery and/or pain related to the musculoskeletal system
* History of eating disorders such as anorexia nervosa, bulimia nervosa were defined as exclusion criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants between the ages of 18-25 who agreed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Bioelectrical Impedance Analysis | two months
  Bioelectrical impedance analysis is a method used to evaluate body composition [30]. Impedance refers to the resistance of tissue to electric current and is inversely proportional to conductivity. For example, components with high specific resistance such as bone and fat tissue make it difficult for electric current to pass, while components with low resistance such as skeletal muscle and visceral organs can easily conduct electric current. This principle forms the basis of bioelectrical impedance analysis [31,32]. Values of < 8.87 kg/m2 in men and < 6.42 kg/m2 in women were considered low muscle mass [9].
  The Tanita BC 401 device will be used in the current study. Participants will be informed before the BIA measurement and will be asked not to drink alcohol for up to 48 hours, not to eat or drink 4 hours before, not to consume tea, coffee and cola for 12 hours before, and not to exercise. In addition, women's measurements will be taken outside of the menstrual period [33,34].
Assessment of Muscle Strength | two months
  Grip strength, will be measured using the JAMAR hand dynamometer and standardized protocol [37]. The JAMAR hand dynamometer is a reliable and most widely used measurement tool for measuring static grip strength [35,38]. Measurements are based on the principle of compressing two parallel bars. The participant is given a position suitable for holding and grip strength and the evaluation is made [38,41]. The needle of the JAMAR Hand Dynamometer can measure up to 90 kg [37,39,42]. The person should sit on a seat without arm support, with the arm in adduction and neutral rotation, the elbow in 90-degree flexion and the forearm in a neutral position [43,44]. The average of three trials for each hand was used to determine general grip strength. Inadequacy in hand grip strength was determined as less than 20 kg for women and less than 30 kg for men [45].
Assessment of Muscle Performance: 4-Meter Walk Test(4-MWT) | two months
  4-Meter Walk Test(4-MWT): (4-MWT) is a walking speed test that evaluates functional limitations and physical performance. (4-MWT) is a widely used test due to its simplicity and high test-retest reliability [46]. Test walking speed is the most commonly used and practical method for evaluating muscle performance in the clinic. A normal value is approximately 3.57 seconds. Additionally, walking speeds of less than 0.8 m/s have been associated with a risk of falling [46,49].
Assessment of Muscle Performance: Sit-to-Stand Test(SST) | two months
  Sit-to-Stand Test(SST): The participant is asked to stand up and sit down completely from a chair for one minute with the arms crossed at chest height from a standard chair height of 45 cm. The number of times the person stands up and sits down completely constitutes the total score [50]. During the test, the participant is seated upright on a chair with their feet touching the floor. The person's arms are crossed in front of their chest. The test is started with the command and the number of times the person gets up completely within 30 seconds is recorded. Only a chair and a stopwatch are required for the test. In the evaluations made for young adults, while for men, results below 15 repetitions in the 30-second sit-to-stand test can be considered as poor performance, this limit is determined as 12 repetitions for women [51].

SECONDARY OUTCOMES:
Assessment of Posture Angles | two months
  The camera, which is placed perpendicular to the floor with a tripod, will be placed 80 cm away from the participant, at the level of the participant's shoulders. The participant is asked to focus on a point at eye level. After taking a lateral photo of the participants while standing, the following posture angles will be calculated using a special software [52,58].
Evaluation of Spinal Muscle Elasticity | two months
  The stiffness and elasticity of the relevant muscles will be evaluated using the MyotonPRO device, which provides information about the stiffness and elasticity of the muscle [59,60]. The participant will be asked to sit on a chair for the assessment. In this way, the participant will be able to reveal his/her completely comfortable position [60]. The relevant points will be marked and the measurement will be carried out perpendicular to this point with MyotonPRO. The measurement will be performed bilaterally on the right and left sides, and the data obtained will be recorded.
Evaluation of The Strength And Endurance of The Spine Stabilization Muscles | two months
  The Stabilizer Pressure Biofeedback Unit will be used to measure the strength with Posterior pelvic tilt movement, isolated Transversus Abdominis strength measurement and Deep Cervical Flexors strength and endurance assessment will be performed using the Stabilizer Pressure Biofeedback Unit [61,62]. The McGill protocol will be used to evaluate core endurance [63].
Measurement of The Strength With The Posterior Pelvic Tilt Movement | two months
  The participant is placed on his back, with the midpoint of the cuff placed on the midpoint of the line connecting both crista iliacae. The manometer valve is closed and the cuff is inflated to a pressure of 40 mm-Hg, and the participant is asked to press his/her waist down without moving his/her head, shoulders and knees, and to wait for 10 seconds without holding his/her breath. The pressure value on the manometer is recorded. The measurement is repeated 3 times with 30-second rest periods, and the maximum value is accepted as the Posterior pelvic tilt muscle strength [64,65].
Transversus Abdominis Strength Measurement | two months
  After the participant is laid face down, the pressure biofeedback unit cuff is placed between the midpoint of the line connecting both spina iliaca anterior superiors and the umbilicus. The participant is asked to breathe comfortably in the abdomen, the valve of the manometer is closed and the cuff is inflated to a pressure of 70 mm-Hg. The participant is asked to pull his abdomen in without moving his spine and pelvis and wait for 10 seconds. The amount of pressure decrease in the manometer is recorded. The measurement is repeated 3 times with 30-second rest periods and the maximum value is recorded as M. transversus abdominis muscle strength[61,66-68].
Endurance Measurement With Deep Cervical Flexor Muscle Strength With Stabilizer | two months
  For measurement, the patient is laid on his/her back on a flat surface. The knees should be bent and the feet should be flat on the floor. The neck is placed in a natural position without a pillow under the head. The stabilizer is placed under the patient's neck, between the occiput and cervical vertebrae. Initially, it is set to 20 mmHg pressure. The patient is instructed to increase the pressure on the stabilizer by slightly pulling the chin in and keeping the head in a neutral position. This movement allows the deep cervical flexor muscles to work actively. The patient gradually increases the pressure to 22 mmHg, 24 mmHg, 26 mmHg, 28 mmHg and 30 mmHg. Each pressure level is held for 10 seconds. If there is no increase in the pressure levels or the patient cannot control the movement, the test is stopped. The value that the error last held for 10 seconds is recorded [69].
Assessment of Core Endurance | two months
  To be assessed using the McGill protocol [63]. Measurements are made using a stopwatch, and results are recorded in seconds. Tests will be terminated when the subject loses position or when the subject says they cannot continue the test [70].
  For the Modified 'Biering-Sorensen' Trunk Extension, the subject is positioned in a prone position with the pelvis, hips, and knees on the bed. The subject is asked to extend their upper body straight forward from the edge of the treatment table.
  For the Trunk Flexors, the subject is positioned with the trunk in 60° flexion, with the knees and hips in 90° flexion. The test is terminated when 60° of trunk flexion is lost.
  For the Prone Bridge, the individual is asked to lie face down, with their elbows flexed, and lift their body up by placing their weight on their forearms and toes. The test is terminated when the position is disrupted.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Orsso CE, Tibaes JRB, Oliveira CLP, Rubin DA, Field CJ, Heymsfield SB, Prado CM, Haqq AM. Low muscle mass and strength in pediatrics patients: Why should we care? Clin Nutr. 2019 Oct;38(5):2002-2015. doi: 10.1016/j.clnu.2019.04.012. Epub 2019 Apr 18. PMID 31031136
- [Background] Clark BC, Manini TM. Functional consequences of sarcopenia and dynapenia in the elderly. Curr Opin Clin Nutr Metab Care. 2010 May;13(3):271-6. doi: 10.1097/MCO.0b013e328337819e. PMID 20154609
- [Background] Manini TM, Clark BC. Dynapenia and aging: an update. J Gerontol A Biol Sci Med Sci. 2012 Jan;67(1):28-40. doi: 10.1093/gerona/glr010. Epub 2011 Mar 28. PMID 21444359
- [Background] Newman AB, Kupelian V, Visser M, Simonsick EM, Goodpaster BH, Kritchevsky SB, Tylavsky FA, Rubin SM, Harris TB. Strength, but not muscle mass, is associated with mortality in the health, aging and body composition study cohort. J Gerontol A Biol Sci Med Sci. 2006 Jan;61(1):72-7. doi: 10.1093/gerona/61.1.72. PMID 16456196
- [Background] Xue QL, Beamer BA, Chaves PH, Guralnik JM, Fried LP. Heterogeneity in rate of decline in grip, hip, and knee strength and the risk of all-cause mortality: the Women's Health and Aging Study II. J Am Geriatr Soc. 2010 Nov;58(11):2076-84. doi: 10.1111/j.1532-5415.2010.03154.x. PMID 21054287
- [Background] Clark BC, Manini TM. What is dynapenia? Nutrition. 2012 May;28(5):495-503. doi: 10.1016/j.nut.2011.12.002. PMID 22469110
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Andreo-Lopez MC, Zarco-Martin MT, Contreras-Bolivar V, Fernandez-Soto ML. Prevalence of Sarcopenia and Dynapenia and Related Clinical Outcomes in Patients with Type 1 Diabetes Mellitus. Nutrients. 2023 Nov 24;15(23):4914. doi: 10.3390/nu15234914. PMID 38068772
- [Background] Ammar A, Brach M, Trabelsi K, Chtourou H, Boukhris O, Masmoudi L, Bouaziz B, Bentlage E, How D, Ahmed M, Muller P, Muller N, Aloui A, Hammouda O, Paineiras-Domingos LL, Braakman-Jansen A, Wrede C, Bastoni S, Pernambuco CS, Mataruna L, Taheri M, Irandoust K, Khacharem A, Bragazzi NL, Chamari K, Glenn JM, Bott NT, Gargouri F, Chaari L, Batatia H, Ali GM, Abdelkarim O, Jarraya M, Abed KE, Souissi N, Van Gemert-Pijnen L, Riemann BL, Riemann L, Moalla W, Gomez-Raja J, Epstein M, Sanderman R, Schulz SV, Jerg A, Al-Horani R, Mansi T, Jmail M, Barbosa F, Ferreira-Santos F, Simunic B, Pisot R, Gaggioli A, Bailey SJ, Steinacker JM, Driss T, Hoekelmann A. Effects of COVID-19 Home Confinement on Eating Behaviour and Physical Activity: Results of the ECLB-COVID19 International Online Survey. Nutrients. 2020 May 28;12(6):1583. doi: 10.3390/nu12061583. PMID 32481594
- [Background] Faulkner JA, Larkin LM, Claflin DR, Brooks SV. Age-related changes in the structure and function of skeletal muscles. Clin Exp Pharmacol Physiol. 2007 Nov;34(11):1091-6. doi: 10.1111/j.1440-1681.2007.04752.x. PMID 17880359
- [Background] Wahlstrom J. Ergonomics, musculoskeletal disorders and computer work. Occup Med (Lond). 2005 May;55(3):168-76. doi: 10.1093/occmed/kqi083. PMID 15857896
- [Background] Callaghan JP, McGill SM. Low back joint loading and kinematics during standing and unsupported sitting. Ergonomics. 2001 Feb 20;44(3):280-94. doi: 10.1080/00140130118276. PMID 11219760
- [Background] Herzog W. Mechanisms of enhanced force production in lengthening (eccentric) muscle contractions. J Appl Physiol (1985). 2014 Jun 1;116(11):1407-17. doi: 10.1152/japplphysiol.00069.2013. Epub 2013 Feb 21. PMID 23429875
- [Background] Rassier DE, MacIntosh BR, Herzog W. Length dependence of active force production in skeletal muscle. J Appl Physiol (1985). 1999 May;86(5):1445-57. doi: 10.1152/jappl.1999.86.5.1445. PMID 10233103
- [Background] Flatters I, Mushtaq F, Hill LJ, Holt RJ, Wilkie RM, Mon-Williams M. The relationship between a child's postural stability and manual dexterity. Exp Brain Res. 2014 Sep;232(9):2907-17. doi: 10.1007/s00221-014-3947-4. Epub 2014 May 14. PMID 24825824
- [Background] Aird L, Samuel D, Stokes M. Quadriceps muscle tone, elasticity and stiffness in older males: reliability and symmetry using the MyotonPRO. Arch Gerontol Geriatr. 2012 Sep-Oct;55(2):e31-9. doi: 10.1016/j.archger.2012.03.005. Epub 2012 Apr 13. PMID 22503549
- [Background] Chuang LL, Wu CY, Lin KC. Reliability, validity, and responsiveness of myotonometric measurement of muscle tone, elasticity, and stiffness in patients with stroke. Arch Phys Med Rehabil. 2012 Mar;93(3):532-40. doi: 10.1016/j.apmr.2011.09.014. Epub 2012 Jan 4. PMID 22222143
- [Background] Conable K, Corneal J, Hambrick T, Marquina N, Zhang J. Investigation of Methods and Styles of Manual Muscle Testing by AK Practitioners. J Chiropr Med. 2005 Winter;4(1):1-10. doi: 10.1016/S0899-3467(07)60106-2. PMID 19674640
- [Background] von Garnier K, Koveker K, Rackwitz B, Kober U, Wilke S, Ewert T, Stucki G. Reliability of a test measuring transversus abdominis muscle recruitment with a pressure biofeedback unit. Physiotherapy. 2009 Mar;95(1):8-14. doi: 10.1016/j.physio.2008.10.003. Epub 2009 Jan 22. PMID 19627680
- [Background] Bohannon R, Gajdosik R, LeVeau BF. Contribution of pelvic and lower limb motion to increases in the angle of passive straight leg raising. Phys Ther. 1985 Apr;65(4):474-6. doi: 10.1093/ptj/65.4.474. PMID 3983239
- [Background] Harris KD, Heer DM, Roy TC, Santos DM, Whitman JM, Wainner RS. Reliability of a measurement of neck flexor muscle endurance. Phys Ther. 2005 Dec;85(12):1349-55. PMID 16305273
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772